CLINICAL TRIAL: NCT04491929
Title: Selective Internal Radiation Therapy With 90Y Resin Micropheres for Refractory Colorectal Cancer Liver Metastases - SIRT - A Translational Feasibility Study
Brief Title: Selective Internal Radiation Therapy With 90Y Resin Micropheres for Refractory Colorectal Cancer Liver Metastases
Acronym: SIRT
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Louise Bach Callesen, Principal Investigator, Aarhus University Hospital
Other Study IDs: 1-10-72-111-20
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Liver Metastasis Colon Cancer
Keywords: Liver metastasis Colon Cancer; Circulating Tumour DNA; Selective Internal Radiation Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational, feasibility study investigating biological aspects in patients with liver metastasis from colorectal cancer undergoing treatment with SIRT, by translational analysis of biological samples.

DETAILED DESCRIPTION:
In this study, the investigators seek to investigate biological aspects in patients with colorectal cancer liver metastasis undergoing treatment with Selective Internal Radiation Therapy, by translational analysis of biological samples.

SIRT will be conducted as per standard procedure at Aarhus University Hospital. Translational blood samples will be drawn pre-treatment and during follow up.

The total cell free DNA level will be quantified in all samples. The samples will be analysed for tumour specific mutations such as the KRAS, BRAF and NRAS oncogenes.

The investigators expect to include up to 30 patients.

This is a purely observational translational study. Results will be analysed in relation to outcome data.

The study is conducted in collaboration with:

Department of Gastroenterology and Hepatology, Aarhus University Hospital Department of Radiology, Aarhus University Hospital Department of Nuclear Medicine, Aarhus University Hospital

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic colorectal adenocarcinoma with liver dominant disease
* Diagnosis of liver metastasis may be made by histo- or cyto-pathology, or by clinical and imaging criteria.
* The Liver metastasis are not eligible for resection, RFA or SBRT
* All patients must be off all chemotherapeutic regimens for 14 days prior to SIRT treatment
* All patients must be off vascular endothelial growth factor inhibitors for 6 weeks prior to SIRT treatment
* Progressive disease, severe intolerance during or following all standard lines of chemo-therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Age 18 years or older
* Able to understand written information
* Consent to samples for translational research

Exclusion Criteria:

* Pretherapeutic work-up procedure with Tc-99m macroaggregated albumin (MAA) scintigraphy showing extrahepatic foci in GI-tract
* Evidence of any detectable Tc-99m macroaggregated albumin deposition in the stomach or duodenum, after application of established angiographic techniques to stop such deposition
* Previous radiation therapy to the lungs and/or to the upper abdomen overlapping with dose to the liver at interventionist´s decision
* Lung shunt greater than 20% or > 30 Gray radiation absorbed dose to the lungs, at estimated by Tc-99m-MAA
* Pregnancy
* Symptomatic lung disease precluding SIRT at interventionist´s decision
* Active uncontrolled infection
* Any pre-treatment laboratory findings within 30 days of treatment demonstrating: alanine aminotransferase level greater than 5 times upper normal limit and/or serum bilirubin greater than 2 mg/dl (>34 umol/l)
* Current or previously evidence of ascites on CT-scan or physical examination
* Tumour volume greater than 50% of liver volume
* Conditions precluding translational samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with metastatic colorectal cancer with chemorefractory liver dominant disease. Patients are found not eligible for surgical resection, RFA or SBRT by a multidisciplinary tumour board (MDT), and considered candidates for SIRT treatment in order to obtain disease control or resectability.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and translational analysis | When 5 patients are included, the blood samples will be analysed for explorative analysis (expected after the first year). In all we expect to include 30 patients if positive results.
  Investigating potential prognostic and predictive markers for efficacy by molecular characteristics and mutational analysis

SECONDARY OUTCOMES:
Response Rate | 6 months
  According to RECIST 1.1
Progression Free Survival | 3 years
Overall Survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Louise B Callesen, Principal Investigator — Experimental Clinical Oncology
Locations (1):
- Department of Oncology, Aarhus University Hospital, Aarhus N, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No